CLINICAL TRIAL: NCT04268238
Title: Pain Control in Dentin Hypersensitivity in Patients With MIH: Study Protocol for a Randomized, Controlled, Clinical Trial
Brief Title: Pain Control in Dentin Hypersensitivity in Patients With MIH
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMI
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Hypersensitivity Dentin
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Study participants and the outcome assessor of sensitivity will be blind to the procedure. However, the researcher who will apply the products is not blind, due to the different forms of clinical manipulation of products.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Experimental): Two weeks before the start of the study, the volunteers will go through a wash out period, where they should only use oral care products donated by the researchers, which should be used until the end of the study. The oral hygiene kit will contain 1 toothbrush (Professional Lab Series, Colgate Palmolive), 1 toothpaste without desensitizing agent, but with fluorine (Elmex) and 1 dental floss (Colgate). Afterwards, this group will receive no treatment. Instead of the sealant, water will be used and the laser will remain with power 0W, that is, there will be no light emission, giving the group the characteristic of the control group, no treatment.
  Interventions: Procedure: Hygiene Guidance
- Sealant group (Experimental): In this group, besides the instructions described in the control group, the teeth that will be sealed will be isolated. 35% phosphoric acid will be applied for 20 seconds and then it will be necessary to wash and dry the tooth surface. Apply a thin layer of PermaSeal (sealant) for 5 seconds to the tooth surface and light curing for 20 seconds.
  Interventions: Procedure: Hygiene Guidance; Procedure: Sealant Application
- Low Level Laser Group (Experimental): In this group, besides the instructions described in the control group, volunteers will receive irradiation with AsGaAl laser, wavelength of 780 nm (Laser XT Therapy, DMC, São Carlos, SP) with fixed power of 100mW, energy density of 35 J/cm2 (considering a spot size of 0.028 cm2 of this equipment), the dose will be 1 J per point. The irradiation will be performed at a cervical, an apical point and another point exactly on the injury, totaling a dose of 3J. Treatment should be performed in 3 sessions with an ideal 72-hour interval between them.
  Interventions: Procedure: Hygiene Guidance; Radiation: Low Level Laser Application
- Low Level Laser + Sealant Group (Experimental): In this group, patients will receive the treatments described in Control group, Sealant group and Low Level Laser Group.
  Interventions: Procedure: Hygiene Guidance; Procedure: Sealant Application; Radiation: Low Level Laser Application

INTERVENTIONS:
Procedure: Hygiene Guidance — Two weeks before the start of the study, the volunteers will go through a wash out period, where they should only use oral care products donated by the researchers, which should be used until the end of the study. The oral hygiene kit will contain 1 toothbrush (Professional Lab Series, Colgate Palmolive), 1 toothpaste without desensitizing agent, but with fluorine (Elmex) and 1 dental floss (Colgate).
Procedure: Sealant Application — Permaseal (Ultradent) is an unloaded resin based on methacrylate and photopolymerizable. The teeth that will be sealed will be isolated. 35% phosphoric acid will be applied for 20 seconds and then it will be necessary to wash and dry the tooth surface. Apply a thin layer of PermaSeal for 5 seconds to the tooth surface and light curing for 20 seconds. After that, it is necessary to evaluate occlusion.
  Arms: Low Level Laser + Sealant Group; Sealant group
Radiation: Low Level Laser Application — Volunteers will receive irradiation with AsGaAl laser, wavelength of 780nm (Laser XT Therapy, DMC, São Carlos, SP) with fixed power of 100mW, density of energy of 35 J/cm2 (considering a spot size of 0.028cm2 of this equipment), the dose will be 1 J per point. Irradiation will be performed at a cervical, an apical point, and another point exactly on the injury, totaling a dose of 3J. Treatment should be performed in 3 sessions with an ideal 72-hour interval between them.
  Arms: Low Level Laser + Sealant Group; Low Level Laser Group

SUMMARY:
This study aims to evaluate the effectiveness of different protocols in controlling dentin hypersensitivity in patients with teeth affected by MIH. The subjects will be randomly designated in four experimental groups, according to different treatments. Pain will be assessed with the visual analog scale (Visual Analogue Scale - VAS), after stimulation with air from the triple syringe and and an exploratory probe at the time of (initial) recruitment, immediately after treatment, after 1 week and 1 month, 3 and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 35 years old;
* Present good general health;
* Present at least one tooth with dentin hypersensitivity reported in the cervical region, which must have a graduated sensitivity equal to or greater than 4 in the VAS scale.

Exclusion Criteria:

* Present active caries lesions or restoration defects in the tooth to be analyzed;
* Present sufficient dentin loss that requires restorative treatment or periodontal surgery;
* Volunteers who underwent any professional desensitizer treatment in the last 6 months;
* Volunteers who used desensitizing pastes in the 3 months;
* Volunteers who were using anti-inflammatory or analgesic drugs at the time of recruitment;
* Volunteers who are pregnant or breastfeeding.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-03-20 (Estimated); Primary Completion 2020-11-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Evaluated by a Visual Analog Scale (VAS) | Baseline, immediately after treatment, 1 week, 1, 3 and 6 months after treatment.
  Pain will be assessed with the visual analogue scale (Visual Analogue Scale - VAS), after stimulation with air from the triple syringe and an explorer probe.